CLINICAL TRIAL: NCT00481598
Title: Non Invasive Assessment of Liver Glycogen Kinetics and ATP Synthesis in Type1 Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landsteiner Institut (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Landsteiner Institute, Landsteiner Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: JDRF Grant Number: 1-2006-74
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: magnet resonance spectroscopy — magnet resonance spectroscopy

SUMMARY:
Patients with Type 1 diabetes (T1DM) suffer from impaired postprandial hepatic glycogen storage and breakdown, if they are under poor glycaemic control. Poor glycogen storage in the liver puts these patients at risk of fasting hypoglycaemia. Amelioration of glycaemic control could improve these abnormalities and thereby reduce the risk of hypoglycaemia in these patients. The "gold standard" technique for the assessment of hepatic glycogen metabolism in humans, 13 C magnetic resonance spectroscopy (13C-MRS), is expensive and limited to a few centers worldwide. Furthermore, treated type 1 diabetic patients exhibit skeletal muscle insulin resistance when treated insufficiently. This condition can also be reversed by improvement of glycaemic control. Recent studies link skeletal muscle insulin resistance to impaired mitochondrial function. Up to date, the impact of glycaemic control on skeletal muscle mitochondrial function has not yet been assessed.

Aim 1 of our project is to establish a new assessment method for glycogen metabolism. This new method is based on oral administration of 2H2O and acetaminophen.

Our second aim is to examine the impact of improvements of glycaemic control on skeletal muscle mitochondrial function in type 1 diabetic patients.

Our third aim is to assess the ATP-synthesis in T1DM.

We will conduct a prospective study on 14 patients with type 1 diabetes and 14 healthy controls.

On the respective study day, participants will be served three standardized meals, blood sugar will be controlled hourly and blood samples will be drawn at timed intervals to determine glucoregulatory hormones, metabolites and enrichments of [6,6-2H2]glucose.

During the night, four 13C-MRS-measurements will be performed in combination with [6,6-2H2]glucose infusion to assess glucose production, glycogen breakdown and gluconeogenesis.

In addition, patients will drink 3g/kg bodyweight 2H2O and acetaminophen will be administered. Thus the new 2H2O-acetaminophen method will be applied simultaneously with the "gold standard" method.

The following morning, mitochondrial function will be assessed in skeletal muscle from unidirectional flux through ATP synthase by 31P MRS.

TIDM patients will be studied twice. First, under conditions of insufficient glycaemic control and the second time after three months of intensified insulin treatment using CSII pumps aiming at optimized metabolic control. Healthy controls will be studied only once.

To assess muscular mitochondrial function in T1DM we will measure ATP synthesis in a calf muscle with magnetic resonance spectroscopy. First, we will conduct a basal measurement. Thereafter, we will start a hyperinsulinaemic euglycemic calmp to stimulate the ATP synthesis and measure again.

This study will provide information on rates of post absorptive glycogen breakdown, gluconeogenesis, and postprandial glycogen storage in the liver and on the skeletal muscle mitochondrial function under conditions of optimized glycaemic control for 3 months.

Finally, this study will demonstrate whether or not poorly controlled type 1 diabetic patients exhibit abnormalities in muscle mitochondrial function and to what extent those alterations can be reversed by optimized glycaemic control. We expect to validate the 2H2O-acetaminophen method, which will provide justification for a broad scale in clinical studies.

DETAILED DESCRIPTION:
Non-Invasive Assessment of Liver Glycogen-Kinetics in Type1 Diabetics

Background:

Hepatic glycogen is the principal short-term reserve for circulating glucose in humans. Up to 50-60% of endogenous glucose production is derived from hepatic glycogenolysis during overnight fasting. In healthy subjects, deprivation of hepatic glycogen by prolonged fasting (60-65 hours) depresses fasting glucose production and plasma glucose levels approach the hypoglycemic range. T1DM were shown to have lower rates of hepatic glycogen synthesis during feeding and lower rates of glycogenolysis during fasting. Thus, this dangerous condition may develop during overnight fasting.

Importantly, defective hepatic glycogen metabolism in T1D can be therapeutically restored, suggesting that measurements of glycogen kinetics could be useful for evaluating both new and existing therapies of glycemic control.

The accepted "gold standard" for hepatic glycogenolysis measurements in humans involves a direct measurement of the natural abundance 13C hepatic glycogen signal using localized 13C NMR on a high-field clinical whole body magnetic resonance system. This method is only available in a handful of clinical research centers around the world.

Our proposed measurement is highly practical and relatively inexpensive since it involves oral administration of a small amount of deuterated water (2H2O) tracer and a standard dose of Acetaminophen. This new method is based on the analysis of deuterium enrichment of urinary glucuronide, which is derived from the glucose moiety of hepatic UDP-glucose, the immediate hexose precursor pool of glycogen synthesis.

To date, there have been no direct comparisons of the 2H2O measurement and clinical 13C MR methods for quantifying rates of fasting glycogenolysis in T1D subjects.

Mitochondrial dysfunction assessed by impaired myocellular ATP synthesis, is associated with insulin resistance in relatives of T2DM, in patients with overt T2DM and T1DM with poor glycemic control. However it is yet unknown to what extend alterations in hyperglycemia contribute to this abnormality. Our hypothesis is that improvement of hyperglycemia in type 1 diabetic patients who do dot suffer from genetically induced insulin resistance, will increase myocellular ATP synthesis. Thus, this study will examine basal myocellular ATP synthetic flux in patients with type 1 diabetes mellitus before and after improvement of glycemic control. In addition, we will perform hyperinsulinaemic euglycemic clamp tests to stimulate mitochondrial ATP synthesis.

Clinical Protocols:

Simultaneous in vivo 13C NMR and 2H2O-glucuronide measurements of hepatic glycogenolysis (Vienna):

A total of 24 subjects consisting of 12 healthy controls and 12 TID patients, first, in insufficient metabolic control (HbA1c 8.5-10.0%) and again after 3 months of intensified insulin treatment using continuous subcutaneous insulin infusion (CSII pump) aiming at optimized metabolic control (HbA1c <7.5%) will be studied following informed consent at the MR Centre-of-Excellence, Medical University of Vienna.

All measurements will either take place in the Hanusch Hospital (Heinrich Collin Straße 30, A-1140 Vienna) or the MR Center-of-Excellence at the General Hospital of Vienna(Lazerettgasse 14, A-1090 Vienna).

For a 24 hour period before the study, T1D patients will be instructed to omit NPH or Zn-insulin and only use regular insulin to control blood glucose concentrations.

On day 1, staring in the Hanusch Hospital, subjects will ingest 3 standard mixed meals (60% CHO, 20% protein and 20% fat; 720kcal, 710kcal and 800kcal) at 08:00, 13:00 and 18.40. The last meal will be served after transferring to the MR-Centre-of-Excellence and the first MR-measurement.

Blood sugar will be controlled hourly and blood samples will be drawn at timed intervals to determine glucoregulatory hormones and metabolites.

Subjects will be transferred periodically to the magnetic resonance spectroscopy unit, where in vivo 13C NMR spectra lasting 1 hour will be performed at 17.30-18.30 (before dinner), 23:30-0:30, 02:00-03:00 and 06:50-07:50. There will be performed an additional 31P NMR measurement to assess the intramyocellular ATP synthesis of the right leg between 05.30-06.30.

At 22:30, a 8-hour primed infusion of [6,6-2H2]glucose will be started. The priming dose of 5 mg/kg will be adjusted according to fasting blood glucose levels and will be followed by a constant infusion of 0.05 mg/kg/min. Plasma samples will be collected twice before the infusion starts and then from 0:30 -0:50, 3:10 - 3:30 and 6:30-6:50 in ten minutes intervals respectively, to quantify enrichment of plasma [6,6-2H2]glucose.

At 23.00, subjects will ingest 2H2O to 0.3% body water and at 03:00, they will ingest 1000 mg Acetaminophen (Paracetamol).

At 6:00 the participants are instructed to void. This Urine will be collected as Urine 1. Between 06:00 and 08:00, Urine will be collected for recovery of Acetaminophen glucuronide (Urine2) at which point the study will finish. The urine will be evaporated, frozen and sent to Coimbra for analysis.

After day one, intensified insulin treatment using continuous subcutaneous insulin infusion (CSII pump) will start. Patients will be re-measured after three month according to the same protocol.

Healthy controls will be examined only once.

ATP-synthesis will be measured on a separate study day. Patients and healthy controls will be admitted to the MR-Centre-of-Excellence at 6:00 a.m. First, there will be a basal measurement of ATP-synthesis. Thereafter, the clamp will be started and conducted for 4 hours. Then, the second 31P NMR measurement will be performed to assess whether ATP synthesis can be stimulated in T1DM patients.

Participants will be released after a meal at 15:00

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus
* HbA1c at the beginning of the trial between 8,5% and 10%
* Age: 18-50 years
* BMI <30 kg/m2 (due to limited MR diameter)
* Normal routine lab tests (blood cell count, kidney, liver, pancreas, thyroid and neuromuscular function)
* Availability within the local area throughout the study
* Ability to understand and sign the consent forms

Exclusion Criteria:

* Current smoking
* Present drug treatment
* Contraindications for MRS studies: claustrophobia and metalliferous implants
* Pregnancy
* HIV or Hepatitis
* acute disease 2 weeks previous to the examination
* Heart disease
* Hypertension (RR>140/95)
* Liver disease
* Kidney disease
* Pulmonary disease
* Thyroid disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
glycogen metabolism, gluconeogenesis, after 3 months of treatment; | August 2008

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Professor Dr., Study Director — Landsteiner Institute
Locations (1):
- Landsteiner Institute for Endocrinology and Metabolic Diseases, Hanusch Hospital Heinrich Collin Straße 30, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kacerovsky M, Brehm A, Chmelik M, Schmid AI, Szendroedi J, Kacerovsky-Bielesz G, Nowotny P, Lettner A, Wolzt M, Jones JG, Roden M. Impaired insulin stimulation of muscular ATP production in patients with type 1 diabetes. J Intern Med. 2011 Feb;269(2):189-99. doi: 10.1111/j.1365-2796.2010.02298.x. PMID 21205021